CLINICAL TRIAL: NCT01100242
Title: Velcade (Bortezomib) and Sorafenib in Unresected or Metastatic Renal Cell Carcinoma
Brief Title: Velcade and Sorafenib in Unresected or Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0812; NCI-2011-02944 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-08

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; metastatic renal cell cancer; kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Bortezomib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: VELCADE and Sorafenib (Experimental): Patients will be given VELCADE® (bortezomib) 1mg/m2 intravenously on days 1,4,8 & 11 and sorafenib at a dosage of 200 mg orally twice per day. One full course is comprised of 21 days.
  Interventions: Drug: Velcade and Sorafenib

INTERVENTIONS:
Drug: Velcade and Sorafenib — Velcade will be administered intravenously; sorafenib will be self-administered on an outpatient basis. At least 2 courses will be administered to each patient unless there is early progression of disease or unacceptable toxicity. Repeated courses may be given to patients who benefit from the treatment (complete or partial remission or stabilization of disease)
  Other Names: velcade; bortezomib; sorafenib

SUMMARY:
This is an open label, non-randomized, single arm phase II study. The primary objective of this study is to investigate the efficacy of combination of sorafenib and VELCADE® (bortezomib). The primary efficacy endpoint is Progression-Free Survival (PFS). The secondary objectives of this study are to:

Assess the response rate of this combination in this patient population and Assess the toxicity of this combination in this patient population

DETAILED DESCRIPTION:
* Pretreatment, a complete history and physical examination to include performance status, weight and concurrent non-malignant disease and therapy will be done before starting treatment. Prior surgery, chemotherapy, and radiotherapy details will be noted.
* Prior to the initiation of treatment, laboratory studies should include a CBC with differential cell count, platelet count, urinalysis, complete metabolic profile, magnesium and electrocardiogram. A baseline imaging study of the tumor will be performed. Other X-rays will be done as clinically indicated.
* Physical examination, performance status and toxicity recording will be done before each course of therapy.
* During the study, patients will be followed with complete blood count (CBC), differential and platelet counts on days 1, 4, 8, and 11. Chemistries will also be performed before each course within a 3 day leeway prior to treatment. Clinical schedules will be considered when scheduling patients for treatment, specimen collection and processing, and specimen shipment.
* Measureable and evaluable disease will be evaluated by the same imaging studies done at baseline and every 2 courses thereafter to determine tumor response.
* For patients on warfarin, International Normalized Ration (INR) testing will be performed prior to the first cycle, weekly during the first cycle, and then prior to day one for subsequent cycles if the INR is in an acceptable range during the first cycle. If the INR has not been in an acceptable range during the first cycle, the INR will be monitored weekly until the value is stable on three consecutive measurements one week apart.
* Since Sorafenib is a competitive inhibitor of cytochrome P450 isoenzyme 3A4 (CYP3A4) patients will be assessed each cycle for medications or changes in diet that would affect CYP3A4 metabolism.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* All patients, 18 years or older with cytologically confirmed clear cell renal with no prior chemotherapy are eligible.
* Patients must have a life expectancy of at least 12 weeks
* Patients must have a Zebroid performance of 0-2
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of > 1500 cells/mm3 and platelet count > 100,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) < two times the upper limit of normal, and adequate renal function as defined by a Serum creatinine < 1.5 x the upper limit of normal.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Patients with non-measurable disease.
* Patients who are unable to take medications orally.
* Patients with resectable renal cell carcinoma
* Patients with a history of Hepatitis B, or Hepatitis C
* Patients known to be Human Immunodeficiency Virus (HIV) positive
* Patients with poorly controlled diabetes mellitus
* Patients with poorly controlled hypertension or hypotension
* Chronic pulmonary disease and a diffusion capacity < 50 %, or a forced vital capacity (FVC) or forced expiratory volume in 1 second (FEV1) of <50%
* Severe renal impairment (Creatinine clearance [CrCL]< 13 ml/min)
* Patients with known malabsorption syndromes.
* Patient has Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol or sorafenib.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 28 days before enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Patients may receive no other concurrent chemotherapy or radiation therapy (XRT) during this trial.
* Patients may not have received XRT within 4 weeks prior to the first treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-04; Primary Completion 2014-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lauer, MD, Principal Investigator — New Mexico Cancer Research Alliance
Locations (3):
- United States (3):
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - The Cancer Center at Presbyterian, Albuquerque, New Mexico
  - Memorial Medical Center- Cancer Center, Las Cruces, New Mexico

REFERENCES:
- [Derived] Rao A, Lauer R. Phase II study of sorafenib and bortezomib for first-line treatment of metastatic or unresectable renal cell carcinoma. Oncologist. 2015 Apr;20(4):370-1. doi: 10.1634/theoncologist.2015-0055. Epub 2015 Mar 16. PMID 25777345
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Groups:
- VELCADE and Sorafenib: VELCADE® (bortezomib) 1mg/m2 intravenously on days 1,4,8 & 11 and sorafenib at 200 mg orally twice per day. One full course is comprised of 21 days.
Period: Overall Study
Arm/Group | VELCADE and Sorafenib
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VELCADE and Sorafenib
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 61 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival will be measured from the beginning of treatment until there is evidence of progressive disease or death from any cause. Progression is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT) or magnetic resonance imaging (MRI): Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 36 weeks
Measure: Median (Full Range); unit: weeks
Groups:
- VELCADE and Sorafenib: VELCADE® (bortezomib) 1mg/m2 intravenously on days 1,4,8 & 11 and sorafenib at 200 mg orally twice per day. One course is comprised of 21 days.
Arm/Group | VELCADE and Sorafenib
Number analyzed (Participants) | 17
weeks | 13.71 [3.9 to 36.0]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Tumor response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT) or magnetic resonance imaging (MRI:) Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Overall response rate (ORR) is the percentage of patients who achieve a CR or PR
Time Frame: 42 days
Measure: Number; unit: percentage of participants
Arm/Group | VELCADE and Sorafenib
Number analyzed (Participants) | 17
percentage of participants
  Complete response (CR) | 0
  Partial response (PR) | 5.9
  Overall response rate (CR + PR) | 5.9

3. Secondary Outcome: Toxicity Profile
Description: Toxicity is assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Toxicity profile is reported as the number of patients who received at least one dose of on-study treatment and experienced a grade 3 or grade 4 adverse event (AE). For a more complete listing of all AEs experienced by patients on study, please see the Adverse Event section.
Time Frame: 42 days
Measure: Number; unit: participants
Arm/Group | VELCADE and Sorafenib
Number analyzed (Participants) | 17
participants
  Abdominal pain | 2
  Anorexia (loss of appetite) | 2
  Dehydration | 1
  Fatigue | 2
  Hand and foot syndrome | 1
  Hemoglobin | 2
  Hyperglycemia | 1
  Hypertension | 1
  Hypoalbuminemia | 3
  Hypokalemia | 1
  Hyponatremia | 5
  Hypophosphatemia | 4
  Lymphopenia | 4
  Pain - Other (All over body) | 1
  Pain in extremity | 1
  Decreased platelets | 1
  Weight loss | 2

ADVERSE EVENTS:
Time Frame: Up to 42 days following last on-study treatment
Arm/Group | VELCADE and Sorafenib
Serious Adverse Events (participants affected / at risk) | 6/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VELCADE and Sorafenib (N=17)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Infection - Other (Infections and infestations) | 1 (2) — Folliculitis due to staphylococcus
Seizure (Nervous system disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pain - other (General disorders) | 1 (1) — Generalized pain all over body required hospitalization
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VELCADE and Sorafenib (N=17)
Allergic reaction (General disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood - Other (Blood and lymphatic system disorders) | 1 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (42)
Neutrophils decreased (Blood and lymphatic system disorders) | 4 (19)
Platelets decreased (Blood and lymphatic system disorders) | 14 (83)
Hypertension (Cardiac disorders) | 6 (7)
Hypotension (Cardiac disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 9 (18)
Fever (General disorders) | 1 (1)
Weight loss (General disorders) | 5 (8)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Decubitus (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 3 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (3)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 7 (11)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (16)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (11)
Taste alteration (Gastrointestinal disorders) | 4 (4)
Voice changes (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Infection, Dental-tooth (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Edema limbs (General disorders) | 5 (6)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alkaline phosphatase increased (Investigations) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Creatinine increased (Investigations) | 11 (26)
Hyperbilirubinemia (Investigations) | 3 (4)
Hypercalcemia (high calcium levels in blood) (Investigations) | 3 (4)
Hyperglycemia (high glucose levels in blood) (Investigations) | 12 (41)
Hyperkalemia (high potassium levels in blood) (Investigations) | 6 (13)
Hypermagnesemia (high magnesium levels in blood) (Investigations) | 2 (2)
Hypoalbuminemia (high albumin levels in blood) (Investigations) | 12 (22)
Hypocalcemia (low calcium levels in blood) (Investigations) | 8 (28)
Hypokalemia (low potassium levels in blood) (Investigations) | 6 (26)
Hypomagnesemia (low magnesium levels in blood) (Investigations) | 3 (6)
Hyponatremia (low sodium levels in blood) (Investigations) | 12 (46)
Hypophosphatemia (low phosphate levels in blood) (Investigations) | 8 (28)
Leukocytes decreased (Blood and lymphatic system disorders) | 6 (56)
Lymphopenia (Blood and lymphatic system disorders) | 7 (95)
Metabolic/Lab - Other (Investigations) | 1 (1) — Elevated lactate dehydrogenase
Prothombin time increased (Investigations) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness - lower limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (7)
Ear, nose and throat examination abnormal (General disorders) | 1 (1)
Abdominal pain (General disorders) | 5 (7)
Back pain (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (2)
Chest wall pain (General disorders) | 1 (1)
External ear pain (General disorders) | 1 (1)
Kidney pain (General disorders) | 1 (1)
Pain - Other (General disorders) | 2 (2)
Pain in extremity (General disorders) | 5 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes